CLINICAL TRIAL: NCT06259617
Title: Influence of Vigorous Physical Activity and Metabolic Parameters on Structure and Function of the Cardiovascular System in Young Athletes - the MuCAYAplus - Study (Munich Cardiovascular Adaptation in Young Athletes Study)
Brief Title: The Munich Cardiovascular Adaptation in Young Athletes Plus Study
Acronym: MuCAYAplus
Status: Recruiting | Type: Observational
Sponsor: Technical University of Munich (Other)
Collaborators: German Research Foundation (Other)
Responsible Party: Sponsor
Other Study IDs: 516547656
Record Dates: First submitted 2024-01-26; First posted 2024-02-14 (Actual); Last update posted 2024-02-14 (Actual); Status verified 2024-02

CONDITIONS: Exercise
Keywords: Adolescents; Children; Exercise; Physical Activity; Vascular adaptation; Cardial adaptation; Carotid Intima-Media-Thickness; Pulse Wave Velocity; Blood pressure; Athletic performance; Nutritional status; Body composition; Biomarkers
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Whole blood, Serum, Blood Plasma
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The aim of the 3-year longitudinal study is to investigate the cardiovascular system's response to training loads in young athletes. For the first time, these parameters will be examined alongside biochemical and metabolic laboratory measures, as well as body composition. The study focuses on the impact of training frequency and intensity, as well as performance, on cardiovascular structure and function.

The following research questions are being investigated:

What structural and functional cardiovascular changes can be observed in young athletes compared to the norm?

What is the relationship between cardiac and vascular parameters depending on the athletic load (training frequency and intensity) as well as athletic performance?

Do cardiac/vascular parameters change over the course of the study, and what role do athletic load (training frequency and intensity) as well as athletic performance play?

What laboratory chemical changes can be observed in young athletes depending on the athletic load (training frequency and intensity) as well as athletic performance?

What connections exist between laboratory chemical parameters and cardiac and vascular parameters in young athletes?

Is there a correlation between structural and functional cardiovascular changes and body composition as well as eating behavior?

ELIGIBILITY:
Inclusion Criteria:

* Participants aged ≥7 and <18 years, presenting for sports medical examination and meeting the criteria mentioned for a period of 3 years
* Athletes participating in competitions, engaging in regular training in a primary sport, being members of a club or association, and training ≥3 hours per week
* The last intensive training must have occurred 12 hours ago to ensure sufficient recovery
* No acute infection, confirmed by a medical examination on the day of testing
* No orthopedic injury, confirmed by a medical examination on the day of testing
* No chronic disease, confirmed by a medical examination on the day of testing
* Clearance for cardiopulmonary stress testing after a medical examination on the day of testing
* Annual participation (1 time per year) in the sports medical examination for 3 years
* Maintaining regular training, training duration ≥3 hours per week, and participation in competitions

Exclusion Criteria:

* Presence of an acute infection, acute orthopedic injury, or chronic disease
* Missing consent from the participant and/or legal guardian

Ages: 7 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Participants aged ≥7 and <18 years, which are participating in athletic competitions, engage in regular training in a primary sport and are members of a club and/or association, with a training load of ≥3 hours per week The participants are recruited at the Pediatric Sports Medicine Outpatient Clinic at the Chair of Preventive Pediatrics. Children and adolescents voluntarily present themselves for sports fitness examinations, either for their competitive activities or as a requirement. These include young athletes who have been examined in previous years or those undergoing a sports fitness examination for the first time.
Sampling Method: Non-Probability Sample
Enrollment: 250 (Estimated)
Dates: Start 2023-12-01 (Actual); Primary Completion 2026-09 (Estimated); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
Vascular stiffness | Once every year over 3 years
  Vascular stiffness of the A. carotis communis, sonographic assessment, result in (%) strain
Peripheral and central blood pressure | Once every year over 3 years
  Assessment via blood pressure cuff, result in (mmHg)
  Pulse Wave Velocity
Left Ventricular internal end diastolic diameter (LVIDd) | Once every year over 3 years
  Echocardiographic assessment, result in (mm)
Left ventricular posterior wall end diastole (LVPWd) | Once every year over 3 years
  Echocardiographic assessment, result in (mm)
Interventricular septum thickness (IVSd) | Once every year over 3 years
  Echocardiographic assessment, result in (mm)
Left ventricular mass (LVM) | Once every year over 3 years
  Echocardiographic assessment, result in (g)
Relative wall thickness (RWT) | Once every year over 3 years
  Echocardiographic assessment, result in (mm)
Ejection fraction (EF) | Once every year over 3 years
  Echocardiographic assessment, result in (%)
Fractional shortening (FS) | Once every year over 3 years
  Echocardiographic assessment, result in (%)
Left ventricular diastolic function (E', E/E', A', E'/A', E-Wave, A-Wave, E/A) | Once every year over 3 years
  Echocardiographic assessment, result in (cm/s)
Left ventricular systolic function (S', S) | Once every year over 3 years
  Echocardiographic assessment, result in (cm/s)
Left Atrial Diameter and Right Atrial Diameter and Diameter/Body Surface Area | Once every year over 3 years
  Echocardiographic assessment, result in (cm)
Left Atrial and Right Atrial Volume/Body Surface Area | Once every year over 3 years
  Echocardiographic assessment, result in (ml/m²)
Left atrial peak longitudinal strain (L-PALS) | Once every year over 3 years
  Echocardiographic assessment, result in (%)
Left atrial peak contraction strain (L-PACS) | Once every year over 3 years
  Echocardiographic assessment, result in (%)
Left atrial total strain | Once every year over 3 years
  Echocardiographic assessment, result in (%)
Right atrial peak longitudinal strain (R-PALS) | Once every year over 3 years
  Echocardiographic assessment, result in (%)
Right atrial peak contraction strain (R-PACS) | Once every year over 3 years
  Echocardiographic assessment, result in (%)
Global longitudinal strain (GLS) | Once every year over 3 years
  Echocardiographic assessment, result in (%)
Intima-Media-Thickness (IMT) | Once every year over 3 years
  Intima-Media-Thickness (IMT) of the A. carotis communis, sonographic assessment, result in (mm)
Peripheral and central pulse pressure | Once every year over 3 years
  Assessment via blood pressure cuff, result in (mmHg)
Pulse Wave Velocity | Once every year over 3 years
  Assessment via blood pressure cuff, result in (ms)

SECONDARY OUTCOMES:
Physical Fitness | Once every year over 3 years
  Spiroergometric measure of VO2max
Nutritional Status | Once every year over 3 years
  Assessment of dietary habits and nutritional status via the validated Healthy Eating Index (HEI).Originally developed in the USA, it was adapted to the German recommendations on food consumption.Higher scores are associated with higher compliance with the official diet recommendations.
Training Frequency | Once every year over 3 years
  Assessment of training frequency via the MoMo activity questionnaire, result in (minutes/week)
Medical history | Once every year over 3 years
  Current illnesses/injuries,Vaccination status, Allergies, Medication, Dietary supplements, Alcohol- and nicotine consumption, Drug use, Energy Drinks, Dietary Habits, Menarche and menstrual cycle in girls Family history of cardiovascular diseases, Unclear deaths, Sudden cardiac death, Marfan syndrome Training history, Symptoms during exercise such as shortness of breath, dizziness/syncope, palpitations or chest pain
Height | Once every year over 3 years
  Measured via Stadiometer, result in (cm)
Weight | Once every year over 3 years
  Measured on scale, result in (kg)
Body-Mass-Index | Once every year over 3 years
  Calculated from Heigt and Weight, result in (kg/m²)
Bodyfat percentage | Once every year over 3 years
  Measured via bioelectric impedance scale, result in (%)
Fat mass | Once every year over 3 years
  Measured via bioelectric impedance scale, result in (kg)
Fat-free mass | Once every year over 3 years
  Measured via bioelectric impedance scale, result in (kg)
Muscle mass | Once every year over 3 years
  Measured via bioelectric impedance scale, result in (kg)
Water content | Once every year over 3 years
  Measured via bioelectric impedance scale, result in (L)
Waist circumference | Once every year over 3 years
  Measured via measuring tape, result in (cm)
Hip circumference | Once every year over 3 years
  Measured via measuring tape, result in (cm)
Sitting height (cm) | Once every year over 3 years
  Measured via Stadiometer, result in (cm)
Erythrocytes | Once every year over 3 years
  Venous blood sampling and laboratory analysis, result in (/pL),
GOT (AST) | Once every year over 3 years
  Venous blood sampling and laboratory analysis, result in (U/L)
GPT (ALT) | Once every year over 3 years
  Venous blood sampling and laboratory analysis, result in (U/L)
GGT | Once every year over 3 years
  Venous blood sampling and laboratory analysis, result in (U/L)
Cholesterol | Once every year over 3 years
  Venous blood sampling and laboratory analysis, result in (mg/dL)
HDL-Cholesterol | Once every year over 3 years
  Venous blood sampling and laboratory analysis, result in (mg/dL)
Non-HDL (calc.) | Once every year over 3 years
  Venous blood sampling and laboratory analysis, result in (mg/dL)
LDL-Cholesterol | Once every year over 3 years
  Venous blood sampling and laboratory analysis, result in (mg/dL)
Creatinine | Once every year over 3 years
  Venous blood sampling and laboratory analysis, result in (mg/dL)
Uric acid | Once every year over 3 years
  Venous blood sampling and laboratory analysis, result in (mg/dL)
hsCRP | Once every year over 3 years
  Venous blood sampling and laboratory analysis, result in (mg/dL)
fT3 | Once every year over 3 years
  Venous blood sampling and laboratory analysis, result in (pg/mL)
Glutathion peroxidase | Once every year over 3 years
  Venous blood sampling and laboratory analysis, result in (U/L)
Superoxide dismutase | Once every year over 3 years
  Venous blood sampling and laboratory analysis, result in (U/mL)
Endothelin-1 | Once every year over 3 years
  Venous blood sampling, blood plasma preparation and laboratory analysis, result in (pg/mL)
Nitric Oxide | Once every year over 3 years
  Venous blood sampling, blood plasma preparation and laboratory analysis, result in (μmol/L)
Ferritin | Once every year over 3 years
  Venous blood sampling, blood plasma preparation and laboratory analysis, result in (ng/mL)
Leptin | Once every year over 3 years
  Venous blood sampling, blood plasma preparation and laboratory analysis, result in (ng/mL)
Training intensity | Once every year over 3 years
  Assessment of training intensity via the MoMo activity questionnaire, result in (metabolic equivalent task-minutes/week)
Hemoglobin | Once every year over 3 years
  Venous blood sampling and laboratory analysis, result in (g/dL)
HBE/MCH | Once every year over 3 years
  Venous blood sampling and laboratory analysis, result in (pg)
MCV | Once every year over 3 years
  Venous blood sampling and laboratory analysis, result in (fL)
Hematocrit | Once every year over 3 years
  Venous blood sampling and laboratory analysis, result in (%)
MCHC | Once every year over 3 years
  Venous blood sampling and laboratory analysis, result in (g/dL)
RDW (Ery) | Once every year over 3 years
  Venous blood sampling and laboratory analysis, result in (%)
Thrombocytes | Once every year over 3 years
  Venous blood sampling and laboratory analysis, result in (Tsnd/µL)
Leukocytes | Once every year over 3 years
  Venous blood sampling and laboratory analysis, result in (/nL)
Heart Rate | Once every year over 3 years
  Assessment via blood pressure cuff, result in (bpm)

CONTACTS AND LOCATIONS:
Overall Officials: Thorsten Schulz, Dr., Principal Investigator — Technical University of Munich
Locations (1):
- Sportmedizinische Ambulanz für Kinder und Jugendliche, München, Bavaria, Germany

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Baumgartner L, Schulz T, Oberhoffer R, Weberruss H. Influence of Vigorous Physical Activity on Structure and Function of the Cardiovascular System in Young Athletes-The MuCAYA-Study. Front Cardiovasc Med. 2019 Oct 9;6:148. doi: 10.3389/fcvm.2019.00148. eCollection 2019. PMID 31649936